CLINICAL TRIAL: NCT00545610
Title: A 12-Month Follow-Up Study to Protocol 24779 (A Double-blind, Prospective, Randomized, Placebo-controlled Study to Determine the Tolerability, Efficacy, Safety, and Dose Range of Intramyocardial Injections of G-CSF Mobilized Auto CD34+ Cells for Reduction of Angina Episodes in Patients With Refractory Chronic Myocardial Ischemia [ACT34-CMI])
Brief Title: ACT34-CMI -- Adult Autologous CD34+ Stem Cells (Follow-Up Study)
Status: Completed | Type: Observational
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 34976
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Test 1 (n=50): 1 x 10^5 (+/-10%) CD34+ cells/kg of body weight
- Test 2 (n=50): 5 x 10^5 (+/-10%) CD34+ cells/kg of body weight
- Placebo (n=50): Saline plus 5% autologous plasma

SUMMARY:
The purpose of this 12-month, observational, follow-up study is to collect additional data (by telephone contact) with which to assess the efficacy, safety, and effects of intramyocardial injections of adult autologous CD34+ cells on quality of life (QoL) in subjects with chronic refractory myocardial ischemia. No treatments will be administered during this study. However, the investigators and other study site personnel and the subjects will remain blinded to the treatment assignments from the core therapeutic study (# 24779) so as to provide a total of 24 months of blinded data.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received treatment with Auto-CD34+ cells or with placebo and who have completed the final study visit (Month 12) of the core therapeutic study 24779
* Subjects who are willing to comply with the specified follow-up evaluations in this study and to provide written informed consent to participate in this study

Ages: 21 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have received treatment with Auto-CD34+ cells (1 x 10^5 (+/-10%) CD34+ cells/kg or 5 x 10^5 (+/-10%) CD34+ cells/kg)or with placebo (saline plus 5% autologous plasma) and who have completed the final study visit (Month 12) of the core therapeutic study 24779
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Long-term safety of intramyocardial injections of Auto-CD34+ cells relative to placebo for reducing the number of angina episodes in subjects with refractory chronic myocardial ischemia over a 12-month follow-up period. | 12 months

SECONDARY OUTCOMES:
Long-term efficacy of Auto-CD34+ cells relative to placebo for reducing the number of angina episodes in subjects with refractory chronic myocardial ischemia and the effects of this treatment on quality of life (QoL) over a 12-month follow-up period | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Caladrius Study Director, Study Director — Lisata Therapeutics, Inc.
Locations (23):
- United States (23):
  - Cardiology, PC, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Scripps Green Hospital / Scripps Clinical Hospital, La Jolla, California
  - Stanford University Hospital and Clinics, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - University of Florida Health Science Center, Jacksonville, Florida
  - Cardiovascular Institute Florida Hospital, Orlando, Florida
  - The Medical Group of St. Joseph´s, Atlanta, Georgia
  - Northwestern University Medical School, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Caritas St. Elizabeth´s Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Cornell University, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Wisconsin Medical School, Madison, Wisconsin
  - Heart Care Associates, LLC, Milwaukee, Wisconsin